CLINICAL TRIAL: NCT02278250
Title: An Open-Label Study of the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Profile of M4344 (Formerly VX-803) as a Single Agent and in Combination With Cytotoxic Chemotherapy in Participants With Advanced Solid Tumors
Brief Title: First in Human Study of M4344 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS201922-0001; VX14-803-001 (Other: Other); 2014-003838-86 (EudraCT Number)
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Results first posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Solid Tumor; Advanced Solid Tumor
Keywords: VX14-803-001; VX-803; M4344; Advanced Solid Tumor; Cytotoxic Chemotherapy; Carboplatin
MeSH Terms: interventions — BID protein, human; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (18):
- Part A: M4344 10 mg BIW (Experimental): Participants received M4344 at a dose of 10 milligrams (mg) orally twice weekly (BIW) until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 10 mg BIW
- Part A: M4344 20 mg BIW (Experimental): Participants received M4344 at a dose of 20 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 20 mg BIW
- Part A: M4344 40 mg BIW (Experimental): Participants received M4344 at a dose of 40 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 40 mg BIW
- Part A: M4344 80 mg BIW (Experimental): Participants received M4344 at a dose of 80 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 80 mg BIW
- Part A: M4344 160 mg BIW (Experimental): Participants received M4344 at a dose of 160 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 160 mg BIW
- Part A: M4344 300 mg BIW (Experimental): Participants received M4344 at a dose of 300 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 300 mg BIW
- Part A: M4344 450 mg BIW (Experimental): Participants received M4344 at a dose of 450 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 450 mg BIW
- Part A: M4344 700 mg BIW (Experimental): Participants received M4344 at a dose of 700 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 700 mg BIW
- Part A: M4344 1050 mg BIW (Experimental): Participants received M4344 at a dose of 1050 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 1050 mg BIW
- Part A: M4344 1200 mg BIW (Experimental): Participants received M4344 at a dose of 1200 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 1200 mg BIW
- Part A2: M4344 100 mg BID (Experimental): Participants received M4344 at a dose of 100 mg orally twice daily (BID) until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 100 mg BID
- Part A2: M4344 150 mg QD (Experimental): Participants received M4344 at a dose of 150 mg orally once daily (QD) until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 150 mg QD
- Part A2: M4344 250 mg QD (Experimental): Participants received M4344 at a dose of 250 mg orally QD until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 250 mg QD
- Part A2: M4344 350 mg QD (Experimental): Participants received M4344 at a dose of 350 mg orally QD until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 350 mg QD
- Part B1: M4344 350 mg + Carboplatin (Experimental): Participants received M4344 at a dose of 350 mg orally on Day 2 and Day 9 in combination with intravenous infusion of Carboplatin at a dose of Area under the concentration versus time curve 5 (AUC5) on Day 1 of 21-day cycle until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 350 mg QD; Drug: Carboplatin
- Part B1: M4344 400 mg + Carboplatin (Experimental): Participants received M4344 at a dose of 400 mg orally on Day 2 and Day 9 in combination with intravenous infusion of Carboplatin at a dose of AUC5 on Day 1 of 21-day cycle until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 400 mg; Drug: Carboplatin
- Part B1: M4344 500 mg + Carboplatin (Experimental): Participants received M4344 at a dose of 500 mg orally on Day 2 and Day 9 in combination with intravenous infusion of Carboplatin at a dose of AUC5 on Day 1 of 21-day cycle until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 500 mg; Drug: Carboplatin
- Part C: M4344 250 mg QD (Experimental): Participants received M4344 at a dose of 250 mg orally QD until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Interventions: Drug: M4344 250 mg QD

INTERVENTIONS:
Drug: M4344 10 mg BIW — Participants received M4344 at a dose of 10 milligrams (mg) orally twice weekly (BIW) until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A: M4344 10 mg BIW
Drug: M4344 20 mg BIW — Participants received M4344 at a dose of 20 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A: M4344 20 mg BIW
Drug: M4344 40 mg BIW — Participants received M4344 at a dose of 40 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A: M4344 40 mg BIW
Drug: M4344 80 mg BIW — Participants received M4344 at a dose of 80 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A: M4344 80 mg BIW
Drug: M4344 160 mg BIW — Participants received M4344 at a dose of 160 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A: M4344 160 mg BIW
Drug: M4344 300 mg BIW — Participants received M4344 at a dose of 300 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A: M4344 300 mg BIW
Drug: M4344 450 mg BIW — Participants received M4344 at a dose of 450 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A: M4344 450 mg BIW
Drug: M4344 700 mg BIW — Participants received M4344 at a dose of 700 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A: M4344 700 mg BIW
Drug: M4344 1050 mg BIW — Participants received M4344 at a dose of 1050 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A: M4344 1050 mg BIW
Drug: M4344 1200 mg BIW — Participants received M4344 at a dose of 1200 mg orally BIW until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A: M4344 1200 mg BIW
Drug: M4344 100 mg BID — Participants received M4344 at a dose of 100 mg orally twice daily (BID) until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A2: M4344 100 mg BID
Drug: M4344 150 mg QD — Participants received M4344 at a dose of 150 mg orally once daily (QD) until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A2: M4344 150 mg QD
Drug: M4344 250 mg QD — Participants received M4344 at a dose of 250 mg orally QD until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A2: M4344 250 mg QD; Part C: M4344 250 mg QD
Drug: M4344 350 mg QD — Participants received M4344 at a dose of 350 mg orally QD until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part A2: M4344 350 mg QD; Part B1: M4344 350 mg + Carboplatin
Drug: M4344 400 mg — Participants received M4344 at a dose of 400 mg orally on Day 2 and Day 9 until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part B1: M4344 400 mg + Carboplatin
Drug: M4344 500 mg — Participants received M4344 at a dose of 500 mg orally on Day 2 and Day 9 until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Other Names: VX-803
  Arms: Part B1: M4344 500 mg + Carboplatin
Drug: Carboplatin — Participants received intravenous infusion of Carboplatin at a dose of Area Under Curve5 (AUC5) on Day 1 of 21-day cycle until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
  Arms: Part B1: M4344 350 mg + Carboplatin; Part B1: M4344 400 mg + Carboplatin; Part B1: M4344 500 mg + Carboplatin

SUMMARY:
The purpose of this study was to evaluate the safety and tolerability of multiple ascending doses of single-agent M4344 administered twice-weekly (BIW), twice daily (BID) or once daily dose schedule in participants with advanced solid tumors. This investigation is a three part study examining M4344 alone and in combination with carboplatin to determine the safety and maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Part A, A2 and A3: Participants with one histologically or cytologically confirmed malignant advanced solid tumor, for which no standard therapy is available which may convey clinical benefit
* Part B1: Participants with one histologically or cytologically confirmed malignant advanced solid tumor, for which no standard therapy is available which may convey clinical benefit and/or participants must have progressed after at least 1 prior chemotherapy regimen in the metastatic setting, and for which carboplatin would be considered standard of care.
* Part C: Participants with 1 histologically or cytologically confirmed malignant advanced solid tumors for which no recommended standard therapy is available (that is, participants who have exhausted all standard of care options according to National Comprehensive Cancer Network [NCCN] Guidance) which may convey clinical benefit, and whose tumor has at least 1 of the following biomarkers as determined by a central trial assay or by an assay with appropriate regulatory status: - C1 or C4: loss-of-function mutations in the gene ARID1A - C2 or C5: loss-of-function mutations in the genes ATRX and/or DAXX - C3 or C6: loss-of-function mutation in the gene ataxia telangiectasia mutated (ATM) - This mandatory biomarker assessment must be conducted during screening on a fresh tumor biopsy (or a biopsy obtained after the end of the previous treatment regimen). If this is not possible for medical reason(s), available archival tumor material can be used (historical data should not be used to confirm biomarker status)
* Measurable disease either according to RECIST criteria (Version 1.1)
* WHO performance status of 0 or 1
* Life expectancy of greater than or equal to (>=)12 weeks
* Hematological and biochemical indices within acceptable ranges at Screening
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Radiotherapy, unless brief course for palliative therapy, endocrine therapy, target-specific therapy, immunotherapy, or chemotherapy during the 4 weeks (6 weeks for nitrosoureas and Mitomycin-C, and 4 weeks for investigational medicinal products) or 4 drug half-lives before first dose of study drug, whichever is greater
* Part B1: More than 6 cycles of prior therapy with carboplatin
* Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the investigator should not exclude the participant
* Part B1: Any known history of Grade 4 thrombocytopenia with any prior chemotherapy regimen
* Brain metastases unless asymptomatic, treated, stable, and not requiring steroids for at least 4 weeks before first dose of study drug
* Female participants who are already pregnant or lactating, or plan to become pregnant within 6 months of the last dose of study drug are excluded. Female participants of childbearing potential must adhere to contraception guidelines. Female participants will be considered to be of nonchildbearing potential if they have undergone surgical hysterectomy or bilateral oophorectomy or have been amenorrheic for over 2 years with a screening serum follicle-stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal females.
* Male participants with partners of childbearing potential must agree to adhere to contraception guidelines. Men with pregnant or lactating partners or partners who plan to become pregnant during the study or within 6 months of the last dose of study drug are excluded.
* Major surgery less than or equal to (<=) 4 weeks before first dose of study drug or incomplete recovery from a prior major surgical procedure
* Serious co-morbid medical conditions, including clinically-significant cardiac disease
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-01-26 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc., a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (16):
- United States (8):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center (MSKCC), New York, New York
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Froedtert & The Medical College of Wisconsin, Wauwatosa, Wisconsin
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Spain (5):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - "Fundacion Jimenez Diaz START Madrid. Oncology Phase I", Madrid
  - START Madrid. Fundacion Jimenez Diaz- Oncologia-Fase I, Madrid
  - "Hospital Clinico Universitario de Valencia Servicio de Hematologia y Oncologia Medica", Valencia
- United Kingdom (2):
  - Sarah Cannon Research Institute UK, London, Greater London
  - Royal Marsden Hospital, Sutton, Surrey

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- [Result] Jo U, Senatorov IS, Zimmermann A, Saha LK, Murai Y, Kim SH, Rajapakse VN, Elloumi F, Takahashi N, Schultz CW, Thomas A, Zenke FT, Pommier Y. Novel and Highly Potent ATR Inhibitor M4344 Kills Cancer Cells With Replication Stress, and Enhances the Chemotherapeutic Activity of Widely Used DNA Damaging Agents. Mol Cancer Ther. 2021 Aug;20(8):1431-1441. doi: 10.1158/1535-7163.MCT-20-1026. Epub 2021 May 27. PMID 34045232
- [Derived] Burris HA, Berlin J, Arkenau T, Cote GM, Lolkema MP, Ferrer-Playan J, Kalapur A, Bolleddula J, Locatelli G, Goddemeier T, Gounaris I, de Bono J. A phase I study of ATR inhibitor gartisertib (M4344) as a single agent and in combination with carboplatin in patients with advanced solid tumours. Br J Cancer. 2024 Apr;130(7):1131-1140. doi: 10.1038/s41416-023-02436-2. Epub 2024 Jan 29. PMID 38287179
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201922-0001
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217341&parentIdentifier=MS201922-0001&attachmentIdentifier=ea28386b-b325-41e6-9020-84aea7f8b7dc&fileName=20220504_MS201922-0001_CT.gov_SAP_Redaction.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was planned to be conducted in multiple parts; Part A, Part A2, Part B1, Part A3 (Dose escalation), Part C1, Part C2, Part C3, Part C4, Part C5 and Part C6 (Dose expansion). On 10 December 2020, the Sponsor decided to discontinue the development of M4344 and stop enrollment of any new participants. Due to the low number of cohorts and participants, data were not summarized per Part (Part C1, C2 and C3). Also, optional Parts A3, C4, C5, and C6 were not conducted.
Period: Overall Study
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin | Part C: M4344 250 mg QD
Started | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 10 | 7 | 7 | 5 | 7 | 7 | 3 | 7 | 6 | 13
Completed | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 10 | 7 | 7 | 5 | 7 | 7 | 3 | 7 | 6 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin | Part C: M4344 250 mg QD | Total
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 10 | 7 | 7 | 5 | 7 | 7 | 3 | 7 | 6 | 13 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 1 | 1 | 1 | 1 | 2 | 8 | 7 | 6 | 5 | 2 | 5 | 4 | 2 | 3 | 5 | 9 | 64
  >=65 years | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 4 | 3 | 1 | 2 | 3 | 2 | 3 | 1 | 4 | 1 | 4 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 8 | 6 | 4 | 3 | 2 | 4 | 2 | 0 | 2 | 3 | 6 | 45
  Male | 1 | 0 | 2 | 0 | 1 | 0 | 4 | 4 | 4 | 3 | 4 | 3 | 3 | 5 | 3 | 5 | 3 | 7 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 9 | 5 | 6 | 4 | 7 | 6 | 2 | 4 | 5 | 12 | 85
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White | 2 | 1 | 2 | 1 | 1 | 1 | 4 | 12 | 8 | 5 | 4 | 2 | 7 | 6 | 2 | 4 | 3 | 12 | 77
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 2 | 0 | 1 | 1 | 3 | 2 | 1 | 17

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal relationship with this treatment. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, regardless if it is considered related to the medicinal product. Serious AE: AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs are defined as AEs that were reported or worsened on or after start of study drug dosing through the Safety Follow-up Visit. TEAEs included both serious TEAEs and non-serious TEAEs.
Time Frame: up to safety follow-up visit (Week 124.9)
Population: The safety analysis set (SAF) included all enrolled participants who received at least 1 dose of study drug (either M4344 or carboplatin (Part B1 only) with the actual amount > 0 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 10 | 7
Participants | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 10 | 7

2. Primary Outcome: Part A: Number of Participants With Grade 3 or 4 (Greater Than [>] 20 Percent [%] of Total) in Laboratory Parameters Based on National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI-CTCAE v4.0)
Description: Laboratory parameters: hematology and chemistry. Blood samples were collected for analysis of following hematology parameters: Hemoglobin, Erythrocytes, mean corpuscular hemoglobin (MCH), MCH concentration, Mean corpuscular volume, Reticulocytes, Platelets, Leukocytes, Eosinophils, Basophils, Neutrophils, Lymphocytes, Monocytes. Blood samples were collected for analysis of following chemistry parameters: Glucose, Blood urea nitrogen/Urea, Creatinine, Sodium, Potassium, Calcium, Chloride, Magnesium, Bicarbonate, Inorganic phosphate, Total bilirubin, Direct bilirubin, Total protein, Albumin, Creatine kinase, Alkaline phosphatase, Aspartate aminotransferase, Alanine aminotransferase, Lactate dehydrogenase, Uric acid, Thyroid stimulating hormone. Number of participants with Grade 3 or 4 (>20% of total) in laboratory parameters were reported as per NCI-CTCAE v4.0 graded from Grade 1 to 5. Grade 1: Mild, Grade 2: Moderate; Grade 3: Severe. Grade 4: Life-threatening and Grade 5: Death.
Time Frame: up to safety follow-up visit (Week 124.9)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 10 | 7
Participants
  Hematology | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 4

3. Primary Outcome: Part A: Number of Participants With Clinically Relevant Findings in Vital Signs
Description: Vital signs included body temperature, heart rate, systolic and diastolic blood pressure and respiration rate. Number of participants with clinically relevant findings in vital signs were reported. Clinical relevance was decided by Investigator.
Time Frame: up to safety follow-up visit (Week 124.9)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 10 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part A: Number of Participants With Clinically Significant Abnormalities in 12-Lead Electrocardiogram (ECGs)
Description: ECG parameters included PR interval, RR interval, QT interval, QRS duration, QTc intervals (derived using Fridericia's correction method) and heart rate. A 12-lead ECG was recorded with the participant in a supine position after a rest of at least 5 minutes using an ECG machine. Clinical significance was decided by investigator. Number of participants with clinically significant abnormalities in 12-Lead ECGs were reported.
Time Frame: up to safety follow-up visit (Week 124.9)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 10 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

5. Primary Outcome: Part A: Maximum Tolerated Dose (MTD) of M4344 Administered Twice Weekly (BIW)
Description: MTD as per NCI-CTCAE v4.0 is defined as highest dose for a given schedule at which there is no more than 1 dose- limiting toxicity (DLT) in 6 participants. DLT: as related/possibly drug-related: Neutropenia Grade (Gr)4 for > 7 days duration/requiring hemopoietic growth factors; Febrile neutropenia; Infection with Gr3/4 neutropenia; Thrombocytopenia Gr3; Thrombocytopenia Gr4 for > 7 days duration/requiring hemopoietic growth factors; Gr3/4 toxicity to organs other than bone marrow; Gr3/4 increase in bilirubin unless increase is due to inhibition of bilirubin glucuronidation; Death due to drug-related complications; Cardiac: QTc prolongation, Gr2/greater ventricular arrhythmia, severe sustained/symptomatic sinus bradycardia, persistent supraventricular arrhythmia, Symptoms suggestive of congestive heart failure, Troponin-T level consistent with myocardial infarction; drug-related toxicity causes interruption of treatment for > 2 weeks.
Time Frame: up to Cycle 1 (each cycle is of 21 days)
Population: Dose Limiting Toxicity (DLT) Evaluable Set: included all enrolled participants who received at least 1 dose of M4344 and either: Experienced a DLT before the end of Cycle 1 or Received at least 80% of scheduled M4344 doses through the end of Cycle 1.
Measure: Number; unit: milligrams (mg)
Groups:
- Part A: M4344: All participants who received escalated oral doses of M4344 (10 mg, 20 mg, 40 mg, 80 mg, 160 mg, 300 mg, 450 mg, 700 mg, 1050 mg and 1200 mg), twice weekly until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
Arm/Group | Part A: M4344
Number analyzed (Participants) | 42
milligrams (mg) | NA — MTD not determined as development focus of the study shifted to daily monotherapy dosing (Part A2).

6. Primary Outcome: Part A2: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: as for outcome 1
Time Frame: up to safety follow-up visit (Week 39)
Population: The SAF included all enrolled participants who received at least 1 dose of study drug (either M4344 or carboplatin (Part B1 only) with the actual amount > 0 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 7 | 5 | 7 | 7
Participants | 7 | 5 | 7 | 7

7. Primary Outcome: Part A2: Number of Participants With Grade 3 or 4 (Greater Than [>] 20 Percent [%] of Total) in Laboratory Parameters Based on National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v5.0)
Description: Laboratory parameters: hematology and chemistry. Blood samples were collected for analysis of following hematology parameters: Hemoglobin, Erythrocytes, mean corpuscular hemoglobin (MCH), MCH concentration, Mean corpuscular volume, Reticulocytes, Platelets, Leukocytes, Eosinophils, Basophils, Neutrophils, Lymphocytes, Monocytes. Blood samples were collected for analysis of following chemistry parameters: Glucose, Blood urea nitrogen/Urea, Creatinine, Sodium, Potassium, Calcium, Chloride, Magnesium, Bicarbonate, Inorganic phosphate, Total bilirubin, Direct bilirubin, Total protein, Albumin, Creatine kinase, Alkaline phosphatase, Aspartate aminotransferase, Alanine aminotransferase, Lactate dehydrogenase, Uric acid, Thyroid stimulating hormone. Number of participants with Grade 3 or 4 (>20% of total) in laboratory parameters were reported as per NCI-CTCAE v5.0 graded from Grade 1 to 5. Grade 1: Mild, Grade 2: Moderate; Grade 3: Severe. Grade 4: Life-threatening and Grade 5: Death.
Time Frame: up to safety follow-up visit (Week 39)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 7 | 5 | 7 | 7
Participants
  Low lymphocytes | 1 | 1 | 2 | 3
  Total Bilirubin | 3 | 2 | 3 | 3
  Aspartate Aminotransferase | 2 | 1 | 0 | 4
  Alanine Aminotransferase | 2 | 2 | 0 | 3

8. Primary Outcome: Part A2: Number of Participants With Clinically Relevant Findings in Vital Signs
Description: Vital signs included body temperature, heart rate, systolic and diastolic blood pressure and respiration rate. Number of participants with clinically relevant findings were reported. Clinical relevance was decided by Investigator.
Time Frame: up to safety follow-up visit (Week 39)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 7 | 5 | 7 | 7
Participants | 0 | 0 | 0 | 0

9. Primary Outcome: Part A2: Number of Participants With Clinically Significant Abnormalities in 12-Lead Electrocardiogram (ECGs)
Description: ECG parameters included PR interval, RR interval, QT interval, QRS duration, QTc intervals (derived using Fridericia's correction method) and heart rate. A 12-lead ECG was recorded with the participant in a supine position after a rest of at least 5 minutes using an ECG machine. Clinical Significance was determined by investigator. Number of participants with clinically significant abnormalities in 12-lead ECGs were reported.
Time Frame: up to safety follow-up visit (Week 39)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 7 | 5 | 7 | 7
Participants | 0 | 0 | 0 | 0

10. Primary Outcome: Part A2: Maximum Tolerated Dose (MTD) of M4344 Administered With a Dose Dense Schedule
Description: MTD as per NCI-CTCAE v5.0 is defined as highest dose for a given schedule at which there is no more than 1 dose- limiting toxicity (DLT) in 6 participants. DLT: as related/possibly drug-related: Neutropenia Grade (Gr)4 for > 7 days duration/requiring hemopoietic growth factors; Febrile neutropenia; Infection with Gr3/4 neutropenia; Thrombocytopenia Gr3; Thrombocytopenia Gr4 for > 7 days duration/requiring hemopoietic growth factors; Gr3/4 toxicity to organs other than bone marrow; Gr3/4 increase in bilirubin unless increase is due to inhibition of bilirubin glucuronidation; Death due to drug-related complications; Cardiac: QTc prolongation, Gr2/greater ventricular arrhythmia, severe sustained/symptomatic sinus bradycardia, persistent supraventricular arrhythmia, Symptoms suggestive of congestive heart failure, Troponin-T level consistent with myocardial infarction; drug-related toxicity causes interruption of treatment for > 2 weeks.
Time Frame: up to Cycle 1 (each cycle is of 21 days)
Population: DLT evaluable set included all enrolled participants who received at least one dose of M4344 and either: Experienced a DLT before the end of Cycle 1 or Received at least 80% of scheduled M4344 doses through the end of Cycle 1.
Measure: Number; unit: mg
Groups:
- Part A2: M4344: All participants who received escalated oral doses of M4344 (100 mg; BID, 150 mg, 250 mg or 350 mg; QD) until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
Arm/Group | Part A2: M4344
Number analyzed (Participants) | 26
mg | 250

11. Primary Outcome: Part B1: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: as for outcome 1
Time Frame: up to Safety follow-up (Week 92.3)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 3 | 7 | 6
Participants | 3 | 7 | 6

12. Primary Outcome: Part B1: Number of Participants With Grade 3 or 4 (Greater Than [>] 20 Percent [%] of Total) in Laboratory Parameters Based on National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI-CTCAE v4.0)
Description: as for outcome 2
Time Frame: up to Safety follow-up (Week 92.3)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 3 | 7 | 6
Participants
  Neutrophils | 1 | 1 | 5
  Platelets | 1 | 3 | 3
  Low hemoglobin | 1 | 4 | 1
  Low Leukocytes | 0 | 1 | 4
  Low lymphocytes | 1 | 3 | 1
  Chemistry | 0 | 0 | 0

13. Primary Outcome: Part B1: Number of Participants With Clinically Relevant Findings in Vital Signs
Description: as for outcome 3
Time Frame: up to Safety follow-up (Week 92.3)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 3 | 7 | 6
Participants | 0 | 0 | 0

14. Primary Outcome: Part B1: Number of Participants With Clinically Significant Abnormalities in 12-Lead Electrocardiogram (ECGs)
Description: as for outcome 9
Time Frame: up to Safety follow-up (Week 92.3)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 3 | 7 | 6
Participants | 0 | 0 | 0

15. Primary Outcome: Part B1: Maximum Tolerated Dose (MTD) of M4344 (Monotherapy) Administered in Combination With Carboplatin
Description: as for outcome 5
Time Frame: up to Cycle 1 (each cycle is of 21 days)
Population: DLT evaluable set included all enrolled participants who received at least one dose of M4344 and either: Experienced a DLT before the end of Cycle 1 or Received Carboplatin dose on Day 1 and M4344 dose on Days 2 and 9.
Measure: Number; unit: mg
Groups:
- Part B1: M4344: All participants who received escalated oral doses of M4344 (350 mg or 400 mg or 500 mg) on Day 2 and Day 9 in combination with intravenous infusion of Carboplatin at a dose of AUC5 on Day 1 of 21-day cycle until disease progression, death, unacceptable toxicity, new anticancer treatment was started, or study withdrawal.
Arm/Group | Part B1: M4344
Number analyzed (Participants) | 16
mg | NA — MTD not determined as development focus of the study shifted to daily monotherapy dosing (Part A2).

16. Primary Outcome: Part C: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment Related AEs According to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Description: AE: any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal relationship with this treatment. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of a medicinal product, regardless if it is considered related to medicinal product. Serious AE: AE that resulted in any of following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs: AEs that were reported/worsened on/after start of study drug dosing through the Safety Follow-up Visit. TEAEs included both serious TEAEs and non-serious TEAEs. Treatment related AEs: reasonably related to the study drug/study treatment. AE could medically (pharmacologically/clinically) be attributed to the study drug/study treatment under study in this clinical study protocol.
Time Frame: up to Safety follow-up (Week 31.1)
Population: The SAF included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: M4344 250 mg QD
Number analyzed (Participants) | 13
Participants
  Participants with TEAEs | 13
  Participants with Treatment related AEs | 13

17. Primary Outcome: Part C: Number of Participants With Grade 3 or 4 (Greater Than [>] 20 Percent [%] of Total) in Laboratory Parameters Based on National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v5.0)
Description: as for outcome 7
Time Frame: up to Safety follow-up (Week 31.1)
Population: The SAF included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: M4344 250 mg QD
Number analyzed (Participants) | 13
Participants
  Low lymphocytes | 8
  Low hemoglobin | 6
  Total Bilirubin | 7
  Aspartate Aminotransferase | 4
  Alanine Aminotransferase | 3

18. Primary Outcome: Part C: Number of Participants With Clinically Relevant Findings in Vital Signs
Description: as for outcome 3
Time Frame: up to Safety follow-up (Week 31.1)
Population: The SAF included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: M4344 250 mg QD
Number analyzed (Participants) | 13
Participants | 0

19. Primary Outcome: Part C: Number of Participants With Clinically Significant Abnormalities in 12-Lead Electrocardiogram (ECGs)
Description: as for outcome 9
Time Frame: up to Safety follow-up (Week 31.1)
Population: The SAF included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: M4344 250 mg QD
Number analyzed (Participants) | 13
Participants | 6

20. Primary Outcome: Part C: Percentage of Participants With Objective Response (OR) According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by the Investigator
Description: OR is defined as the confirmed assessment of best overall response of complete response (CR) or partial response (PR). CR is defined as disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions.
Time Frame: Time from first dose of study treatment up to 6.4 years
Population: Full Analysis Set (FAS) included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part C: M4344 250 mg QD
Number analyzed (Participants) | 13
percentage of participants | 0.0 [0.0 to 20.6]

21. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) of M4344
Description: Cmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: The Pharmacokinetic Analysis Set (PAS) included all enrolled participants who received at least one dose of M4344 with the actual amount > 0 mg and provide at least one measurable post-dose concentration. Participants were analyzed according to the actual treatment they received. Here, "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 10 | 7
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 376 (64.2) | 516 (83.6) | 395 (73.2) | 576 (79.9)
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 2 | 3 | 7 | 6 | 3
  Cycle 1 Day 8 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 342 (136.6) | 675 (65.7) | 328 (313.1) | 486 (23.8)

22. Secondary Outcome: Part A: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of M4344
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: The PAS included all enrolled participants who received at least one dose of M4344 with the actual amount > 0 mg and provide at least one measurable post-dose concentration. Participants were analyzed according to the actual treatment they received. Here, "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 10 | 7
nanogram*hour per milliliter (ng*h/mL)
  Cycle 1 Day 1 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 948 (56.4) | 1830 (102.0) | 1390 (64.5) | 2220 (105.9)
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 2 | 3 | 7 | 6 | 3
  Cycle 1 Day 8 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 809 (96.6) | 2670 (91.2) | 1550 (295.1) | 1880 (74.0)

23. Secondary Outcome: Part A: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of M4344
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLOQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Cycle 1 Day 1 (each cycle is of 21 days)
Population: The Pharmacokinetic Analysis Set (PAS) included all enrolled participants who received at least one dose of M4344 with the actual amount > 0 mg and provide at least one measurable post-dose concentration. Participants were analyzed according to the actual treatment they received. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 10 | 6 | 3
ng*h/mL | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 971 (53.6) | 1710 (92.5) | 1760 (122.3) | 1540 (128.9)

24. Secondary Outcome: Part A: Time to Reach Maximum Plasma Concentration (Tmax) of M4344
Description: Tmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: as for outcome 22
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 10 | 7
hours
  Cycle 1 Day 1 | NA [NA to NA] — Median and Full range were not to be calculated if fewer than 3 participants have reportable parameter values. | NA [NA to NA] — Median and Full range were not to be calculated if fewer than 3 participants have reportable parameter values. | NA [NA to NA] — Median and Full range were not to be calculated if fewer than 3 participants have reportable parameter values. | NA [NA to NA] — Median and Full range were not to be calculated if fewer than 3 participants have reportable parameter values. | NA [NA to NA] — Median and Full range were not to be calculated if fewer than 3 participants have reportable parameter values. | NA [NA to NA] — Median and Full range were not to be calculated if fewer than 3 participants have reportable parameter values. | 1.51 [0.663 to 2.15] | 2.00 [0.533 to 8.00] | 2.06 [1.50 to 4.00] | 3.07 [1.50 to 4.07]
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 2 | 3 | 7 | 6 | 3
  Cycle 1 Day 8 | NA [NA to NA] — Median and Full range were not to be calculated if fewer than 3 participants have reportable parameter values. | NA [NA to NA] — Median and Full range were not to be calculated if fewer than 3 participants have reportable parameter values. | NA [NA to NA] — Median and Full range were not to be calculated if fewer than 3 participants have reportable parameter values. | NA [NA to NA] — Median and Full range were not to be calculated if fewer than 3 participants have reportable parameter values. | NA [NA to NA] — Median and Full range were not to be calculated if fewer than 3 participants have reportable parameter values. | NA [NA to NA] — Median and Full range were not to be calculated if fewer than 3 participants have reportable parameter values. | 1.22 [1.05 to 1.50] | 2.00 [1.57 to 3.95] | 4.00 [1.52 to 8.05] | 3.95 [3.00 to 4.00]

25. Secondary Outcome: Part A: Terminal Elimination Half-Life (T1/2) of M4344
Description: Elimination Half Life (T1/2) was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half. T1/2 was calculated by natural log 2 divided by Lambda z. Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: The PAS included all enrolled participants who received at least one dose of M4344 with the actual amount > 0 mg and provide at least one measurable post-dose concentration. Participants were analyzed according to the actual treatment they received. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 10 | 6 | 3
hours
  Cycle 1 Day 1 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 2.22 (99.0) | 3.33 (42.3) | 4.61 (65.2) | 3.60 (39.9)
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 2 | 3 | 6 | 2 | 0
  Cycle 1 Day 8 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 2.19 (220.1) | 3.11 (64.2) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. |

26. Secondary Outcome: Part A: Apparent Clearance (CL/f) of M4344
Description: CL/f was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. CL/f was calculated as Dose/AUC0-inf, where AUC0-inf was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. AUC0-inf was calculated as AUC0-t + Clast pred/Lambda Z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the lower limit of quantification (LLQ) and Lambda Z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 10 | 6 | 3
liter per hour
  Cycle 1 Day 1 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 464 (53.6) | 409 (92.5) | 597 (122.3) | 781 (128.9)
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 2 | 3 | 6 | 2 | 0
  Cycle 1 Day 8 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 513 (78.2) | 221 (114.3) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. |

27. Secondary Outcome: Part A: Apparent Volume of Distribution During Terminal Phase (Vz/f) of M4344
Description: Vz/f: the distribution of a study drug between plasma and the rest of the body after oral dosing. For single dose Vz/f = Dose/(AUC0-inf*Lambda Z), where AUC0-inf = (AUC0-t + Clast pred/Lambda Z). Clastpred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLOQ and Lambda Z = the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 10 | 6 | 3
liters
  Cycle 1 Day 1 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 1480 (187.9) | 1960 (116.0) | 3970 (95.8) | 4060 (211.6)
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 2 | 3 | 6 | 2 | 0
  Cycle 1 Day 8 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 1620 (716.8) | 993 (59.6) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. |

28. Secondary Outcome: Part A: Accumulation Ratio for Maximum Observed Plasma Concentration (Racc [Cmax]) of M4344
Description: Accumulation ratio of Cmax was calculated as Cmax, after dosing on Day 8 divided by Cmax, after dosing on Day 1 of Cycle 1.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: The PAS included all enrolled participants who received at least one dose of M4344 with the actual amount > 0 mg and provide at least one measurable post-dose concentration. Participants were analyzed according to the actual treatment they received. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 2 | 3 | 7 | 6 | 3
ratio | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 0.988 (37.9) | 1.19 (67.5) | 1.01 (163.2) | 1.55 (17.4)

29. Secondary Outcome: Part A: Accumulation Ratio for Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (Racc [AUC0-t]) of M4344
Description: Accumulation ratio of AUC0-t was calculated as AUC0-t, after dosing on Day 8 divided by AUC0-t, after dosing on Day 1 of Cycle 1.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 2 | 3 | 7 | 6 | 3
ratio | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 0.955 (23.7) | 1.46 (77.8) | 1.36 (163.7) | 1.89 (33.6)

30. Secondary Outcome: Part A: Dose Normalized Maximum Observed Plasma Concentration (Cmax/Dose) of M4344
Description: Dose normalized was calculated as Cmax obtained directly from the concentration versus time curve divided by dose. Cmax/dose was measured in nanogram per milliliter per milligram (ng/mL/mg).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 10 | 7
ng/mL/mg
  Cycle 1 Day 1 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 0.835 (64.2) | 0.738 (83.6) | 0.376 (73.2) | 0.480 (79.9)
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 3 | 7 | 6 | 3
  Cycle 1 Day 8 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 0.760 (136.6) | 0.964 (65.7) | 0.312 (313.1) | 0.405 (23.8)

31. Secondary Outcome: Part A: Dose Normalized Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-t/Dose) of M4344
Description: AUC0-t/Dose was defined as AUC from time of dosing to the time of the last measurable concentration divided by dose. AUC0-t/dose was measured in nanogram*hour per milliliter per milligram (ng*h/mL/mg).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 12 | 10 | 7
ng*h/mL/mg
  Cycle 1 Day 1 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 2.11 (56.4) | 2.61 (102.0) | 1.32 (64.5) | 1.85 (105.9)
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 3 | 7 | 6 | 3
  Cycle 1 Day 8 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 1.80 (96.6) | 3.82 (91.2) | 1.47 (295.1) | 1.57 (74.0)

32. Secondary Outcome: Part A: Dose Normalized Area Under the Concentration-Time Curve Over Entire Dosing Time Period From Time Zero Extrapolated to Infinity (AUC0-inf/Dose) of M4344
Description: AUC0-inf/Dose was defined as AUC extrapolated to infinity divided by dose.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8, and 24 hours post-dose on Cycle 1 Day 1 (each cycle is of 21 days)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 4 | 10 | 6 | 3
ng*h/mL/mg | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 2.16 (53.6) | 2.45 (92.5) | 1.68 (122.3) | 1.28 (128.9)

33. Secondary Outcome: Part A: Percentage of Participants With Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: The OR was defined as the confirmed assessment of best overall response (BOR) of partial response (PR),or complete response (CR) according to RECIST v1.1. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in sum of longest diameter (SLD) of all lesions.
Time Frame: Time from first dose of study treatment up to 4.3 years
Population: Full analysis set (FAS): all enrolled participants who satisfy all of the following criteria: received at least 1 dose of study drug with the actual amount > 0 mg; have a baseline scan with a measurable target lesion (sum of diameters of all target lesions > 0 mm) and have at least 1 disease assessment on treatment with a measurable target lesion (sum of diameters of all target lesions >= 0 mm); or subjects who have discontinued the study due to either progressive disease or death.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 6 | 7 | 4
percentage of participants | 0.0 [0.0 to 95.0] | 0.0 [0.0 to 95.0] | 0.0 [0.0 to 95.0] | 0.0 [0.0 to 95.0] | 0.0 [0.0 to 95.0] | 0.0 [0.0 to 95.0] | 0.0 [0.0 to 63.2] | 0.0 [0.0 to 39.3] | 0.0 [0.0 to 34.8] | 0.0 [0.0 to 52.7]

34. Secondary Outcome: Part A: Number of Participants With Stable Disease (SD) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: SD is defined as neither sufficient increase to qualify for progression disease (PD) nor sufficient shrinkage to qualify for partial response (PR). PR: at least 30 percent (%) reduction from baseline in sum of longest diameter (SLD) of all lesions. PD: at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from first dose of study treatment up to 4.3 years
Population: FAS: all enrolled participants who satisfy all of the following criteria: received at least 1 dose of study drug with the actual amount > 0 mg; have a baseline scan with a measurable target lesion (sum of diameters of all target lesions > 0 mm) and have at least 1 disease assessment on treatment with a measurable target lesion (sum of diameters of all target lesions >= 0 mm); or subjects who have discontinued the study due to either progressive disease or death.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 6 | 7 | 4
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1

35. Secondary Outcome: Part A2: Maximum Observed Plasma Concentration (Cmax) of M4344
Description: Cmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: The PAS included all enrolled participants who received at least one dose of M4344 with the actual amount > 0 mg and provide at least one measurable post-dose concentration. Participants were analyzed according to the actual treatment they received. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 6 | 5 | 7 | 7
ng/mL
  Cycle 1 Day 1 | 111 (40.3) | 124 (392.2) | 517 (78.3) | 265 (152.7)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 7 | 2
  Cycle 1 Day 8 | 114 (32.3) | 244 (59.3) | 379 (88.9) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values.

36. Secondary Outcome: Part A2: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of M4344
Description: as for outcome 23
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose on Cycle 1 Day 1 (each cycle is of 21 days)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 6 | 5 | 6 | 7
ng*h/mL | 217 (44.2) | 436 (127.4) | 1210 (95.0) | 680 (144.1)

37. Secondary Outcome: Part A2: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of M4344
Description: as for outcome 22
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 (in BID arms), 24 hours post-dose (in QD arms) on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 6 | 5 | 7 | 7
ng*h/mL
  Cycle 1 Day 1 | 216 (43.2) | 414 (142.9) | 1230 (86.1) | 703 (142.7)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 7 | 2
  Cycle 1 Day 8 | 236 (55.4) | 627 (58.9) | 829 (101.4) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values.

38. Secondary Outcome: Part A2: Time to Reach Maximum Plasma Concentration (Tmax) of M4344
Description: Tmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: as for outcome 25
Measure: Median (Full Range); unit: hours
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 6 | 5 | 7 | 7
hours
  Cycle 1 Day 1 | 1.45 [0.517 to 2.00] | 1.62 [0.467 to 2.07] | 1.50 [0.500 to 2.00] | 1.10 [0.683 to 3.02]
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 7 | 2
  Cycle 1 Day 8 | 1.03 [1.00 to 1.43] | 1.28 [0.500 to 2.00] | 1.50 [0.500 to 1.95] | NA [NA to NA] — Median and Full range were not to be calculated if fewer than 3 participants have reportable parameter values.

39. Secondary Outcome: Part A2: Terminal Elimination Half-Life (T1/2) of M4344
Description: as for outcome 25
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 6 | 5 | 7 | 7
hours
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 5 | 6 | 7
  Cycle 1 Day 1 | 1.32 (27.1) | 2.47 (165.9) | 1.74 (58.8) | 2.37 (60.9)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 7 | 2
  Cycle 1 Day 8 | 1.36 (58.7) | 1.31 (28.9) | 1.31 (18.7) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values.

40. Secondary Outcome: Part A2: Apparent Clearance (CL/f) of M4344
Description: as for outcome 26
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 6 | 5 | 7 | 7
liter per hour
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 5 | 6 | 7
  Cycle 1 Day 1 | 461 (44.2) | 344 (127.4) | 207 (95.0) | 515 (144.1)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 7 | 2
  Cycle 1 Day 8 | 424 (55.4) | 239 (58.9) | 302 (101.4) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values.

41. Secondary Outcome: Part A2: Apparent Volume of Distribution During Terminal Phase (Vz/f) of M4344
Description: as for outcome 27
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose on Cycle 1 Day 1 (each cycle is of 21 days)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 6 | 5 | 6 | 7
liters | 876 (36.3) | 1220 (661.7) | 519 (191.1) | 1760 (214.7)

42. Secondary Outcome: Part A2: Accumulation Ratio for Maximum Observed Plasma Concentration (Racc [Cmax]) of M4344
Description: as for outcome 28
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 3 | 4 | 7 | 2
ratio | 1.08 (47.5) | 2.26 (245.2) | 0.733 (92.1) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values.

43. Secondary Outcome: Part A2: Accumulation Ratio for Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (Racc [AUC0-t]) of M4344
Description: as for outcome 29
Time Frame: as for outcome 37
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 3 | 4 | 7 | 2
ratio | 1.00 (55.3) | 1.42 (142.4) | 0.672 (90.7) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values.

44. Secondary Outcome: Part A2: Accumulation Ratio for Area Under the Plasma Concentration Time Curve (Racc [AUC]) of M4344
Description: Accumulation ratio of AUC was calculated as AUC, after dosing on Day 8 divided by AUC, after dosing on Day 1 of Cycle 1.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 3 | 4 | 7 | 2
ratio | 0.997 (55.7) | 1.32 (133.5) | 0.676 (88.4) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values.

45. Secondary Outcome: Part A2: Dose Normalized Maximum Observed Plasma Concentration (Cmax/Dose) of M4344
Description: as for outcome 30
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose on Day 1 and Day 8 of Cycle 1 (each cycle is of 21 days)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 6 | 5 | 7 | 7
ng/mL/mg
  Cycle 1 Day 1 | 1.11 (40.3) | 0.829 (392.2) | 2.07 (78.3) | 0.758 (152.7)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 7 | 2
  Cycle 1 Day 8 | 1.14 (32.3) | 1.63 (59.3) | 1.52 (88.9) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values.

46. Secondary Outcome: Part A2: Dose Normalized Area Under the Concentration-Time Curve Over Entire Dosing Time Period From Time Zero Extrapolated to Infinity (AUC0-inf/Dose) of M4344
Description: AUC0-inf/Dose was defined as AUC extrapolated to infinity divided by dose. AUC0-inf/Dose was measured in nanogram*hour per milliliter per milligram (ng*h/mL/mg).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose on Cycle 1 Day 1 (each cycle is of 21 days)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 6 | 5 | 6 | 7
ng*h/mL/mg | 2.17 (44.2) | 2.91 (127.4) | 4.84 (95.0) | 1.94 (144.1)

47. Secondary Outcome: Part A2: Dose Normalized Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-t/Dose) of M4344
Description: AUC0-t/Dose was defined as AUC from time of dosing to the time of the last measurable concentration divided by dose.
Time Frame: as for outcome 37
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 6 | 5 | 7 | 7
ng*h/mL/mg
  Cycle 1 Day 1 | 2.16 (43.2) | 2.76 (142.9) | 4.93 (86.1) | 2.01 (142.7)
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 7 | 2
  Cycle 1 Day 8 | 2.36 (55.4) | 4.18 (58.9) | 3.32 (101.4) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values.

48. Secondary Outcome: Part A2: Number of Participants With Stable Disease (SD) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: as for outcome 34
Time Frame: Time from first dose of study treatment up to 6.2 years
Population: FAS is defined as all enrolled participants who received at least 1 dose of study drug, have a baseline scan, and received at least one disease assessment while on treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 7 | 4 | 7 | 5
Participants | 1 | 1 | 4 | 2

49. Secondary Outcome: Part A2: Percentage of Participants With Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: as for outcome 33
Time Frame: Time from first dose of study treatment up to 6.2 years
Population: as for outcome 48
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD
Number analyzed (Participants) | 7 | 4 | 7 | 5
percentage of participants | 0.0 [0.0 to 34.8] | 0.0 [0.0 to 52.7] | 0.0 [0.0 to 34.8] | 0.0 [0.0 to 45.1]

50. Secondary Outcome: Part B1: Maximum Observed Plasma Concentration (Cmax) of M4344
Description: Cmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: The PAS included all enrolled participants who received at least one dose of M4344 with the actual amount > 0 mg and provide at least one measurable post-dose concentration. Participants were analyzed according to the actual treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 3 | 7 | 6
ng/mL | 309 (78.1) | 114 (191.6) | 367 (89.8)

51. Secondary Outcome: Part B1: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of M4344
Description: as for outcome 22
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 50
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 3 | 7 | 6
ng*h/mL | 392 (101.8) | 268 (179.6) | 1450 (115.6)

52. Secondary Outcome: Part B1: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of M4344
Description: as for outcome 23
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 2 | 4 | 3
ng*h/mL | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 368 (147.3) | 2570 (124.3)

53. Secondary Outcome: Part B1:Time to Reach Maximum Plasma Concentration (Tmax) of M4344
Description: Tmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 50
Measure: Median (Full Range); unit: hours
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 3 | 7 | 6
hours | 1.52 [0.900 to 2.00] | 1.50 [0.500 to 8.02] | 1.96 [1.00 to 3.00]

54. Secondary Outcome: Part B1: Terminal Elimination Half-Life (T1/2) of M4344
Description: as for outcome 25
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 2 | 4 | 3
hours | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 1.03 (23.6) | 3.77 (59.1)

55. Secondary Outcome: Part B1: Apparent Clearance (CL/f) of M4344
Description: as for outcome 26
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 2 | 4 | 3
liter per hour | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 1090 (147.3) | 194 (124.3)

56. Secondary Outcome: Part B1: Apparent Volume of Distribution During Terminal Phase (Vz/f) of M4344
Description: as for outcome 27
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 2 | 4 | 3
liters | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 1620 (155.5) | 1060 (45.1)

57. Secondary Outcome: Part B1: Dose Normalized Maximum Observed Plasma Concentration (Cmax/Dose) of M4344
Description: Dose normalized was calculated as Cmax obtained directly from the concentration versus time curve divided by dose.
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 50
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 3 | 7 | 6
ng/mL/mg | 0.884 (78.1) | 0.286 (191.6) | 0.735 (89.8)

58. Secondary Outcome: Part B1: Dose Normalized Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-t/Dose) of M4344
Description: AUC0-t/Dose was defined as AUC from time of dosing to the time of the last measurable concentration divided by dose.
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 50
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 3 | 7 | 6
ng*h/mL/mg | 1.12 (101.8) | 0.669 (179.6) | 2.90 (115.6)

59. Secondary Outcome: Part B1: Dose Normalized Area Under the Concentration-Time Curve Over Entire Dosing Time Period From Time Zero Extrapolated to Infinity (AUC0-inf/Dose) of M4344
Description: AUC0-inf/Dose was defined as AUC extrapolated to infinity divided by dose.
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours post-dose on Cycle 1 Day 2 (each cycle is of 21 days)
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 2 | 4 | 3
ng*h/mL/mg | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not to be calculated if fewer than 3 participants have reportable parameter values. | 0.920 (147.3) | 5.15 (124.3)

60. Secondary Outcome: Part B1: Percentage of Participants With Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: as for outcome 33
Time Frame: Time from first dose of study treatment up to 5.2 years
Population: FAS is defined as all enrolled participants who received at least 1 dose of study treatment, have a baseline scan with a measurable target lesion, and at least one on-treatment disease assessment or have discontinued the study due to either progressive disease or death.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin
Number analyzed (Participants) | 3 | 7 | 6
percentage of participants | 0.0 [0.0 to 63.2] | 14.3 [0.7 to 52.1] | 0.0 [0.0 to 39.3]

61. Secondary Outcome: Part C: Number of Participants With Confirmed Best Overall Response (BOR) as Per Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1
Description: Confirmed BOR is defined as best response of any of complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) recorded from the treatment start date until documented disease progression. CR: Disappearance of all evidence of target/non-target lesions. PR: At least 30%reduction from baseline in sum of longest diameter (SLD) of all lesions. SD: Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD: at least a 20% increase in SLD, taking as reference smallest SLD recorded from baseline/appearance of 1or more new lesions and unequivocal progression of non-target lesions.
Time Frame: Time from first dose of study treatment up to 6.4 years
Population: FAS included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: M4344 250 mg QD
Number analyzed (Participants) | 13
Participants
  Complete response (CR) | 0
  Partial response (PR) | 0
  Stable disease (SD) | 3
  Progressive disease (PD) | 8
  Non-CR/Non-PD | 0
  Non-evaluable | 2

62. Secondary Outcome: Part C: Progression-Free Survival (PFS) as Per Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1 as Assessed by Investigator
Description: PFS is defined as the time from start of study treatment to progression disease (PD) or death. PD: at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Time from first dose of study treatment up to 6.4 years
Population: FAS included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part C: M4344 250 mg QD
Number analyzed (Participants) | 13
months | 1.6 [0.8 to 2.1]

63. Secondary Outcome: Part C: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator
Description: DOR was defined for participants with confirmed response, as the time from first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from first documentation of objective response, assessed up to 6.4 years
Population: As per planned analysis, DoR was not analyzed due to the small number of participants and the low likelihood that any participant would experience an objective response.
Arm/Group | Part C: M4344 250 mg QD
Number analyzed (Participants) | 0

64. Secondary Outcome: Part C: Overall Survival (OS)
Description: OS was defined as the time from treatment start to the date of death due to any cause. The participants who were still alive at the time of data analysis or who were lost to follow-up OS time was censored at the last recorded date. OS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Time from first dose of study treatment up to 6.4 years
Population: FAS included all participants who received at least one dose of study drug. The summarized data was not available for these arms therefore individual data was presented. Here, "Overall Number of Participants" signifies those participants who were evaluable for this outcome measure and "number analyzed" = specific participants evaluated in the arm.
Measure: Number; unit: months
Arm/Group | Part C: M4344 250 mg QD
Number analyzed (Participants) | 6
months
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 1.91
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 0.79
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 1.61
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | 3.98
  Participant 5: number analyzed (Participants) | 1
  Participant 5 | 2.53
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | 2.63

65. Secondary Outcome: Part C: Maximum Observed Plasma Concentration (Cmax) of M4344
Description: Cmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose up to 2 hours post-dose on Cycle 1 Day 1; Pre-dose up to 1 hours post-dose on Cycle 1 Day 8 and Cycle 1 Day 15 (each cycle is of 21 days)
Population: As per changes in planned analysis, the outcome measures related to pharmacokinetic parameters were not assessed for Part C.
Arm/Group | Part C: M4344 250 mg QD
Number analyzed (Participants) | 0

66. Secondary Outcome: Part C: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of M4344
Description: as for outcome 22
Time Frame: as for outcome 65
Population: as for outcome 65
Arm/Group | Part C: M4344 250 mg QD
Number analyzed (Participants) | 0

67. Secondary Outcome: Part C: Time to Reach Maximum Plasma Concentration (Tmax) of M4344
Description: Tmax was obtained directly from the plasma concentration versus time curve.
Time Frame: as for outcome 65
Population: as for outcome 65
Arm/Group | Part C: M4344 250 mg QD
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Part A: up to Safety follow-up (Week 124.9), Part A2: up to Safety follow-up ( Week 39), Part B1: up to Safety follow-up (Week 92.3) and Part C: up to Safety follow-up (Week 31.1)
Description: Part A, A2 and B1: The SAF included all enrolled participants who received at least 1 dose of study drug (either M4344 or carboplatin (Part B1 only) with the actual amount > 0 mg. Part C: The SAF included all participants who received at least one dose of study drug. For Part A and B: MedDRA version 23.0 and for Part A2 and C: MedDRA version 24.0.
Arm/Group | Part A: M4344 10 mg BIW | Part A: M4344 20 mg BIW | Part A: M4344 40 mg BIW | Part A: M4344 80 mg BIW | Part A: M4344 160 mg BIW | Part A: M4344 300 mg BIW | Part A: M4344 450 mg BIW | Part A: M4344 700 mg BIW | Part A: M4344 1050 mg BIW | Part A: M4344 1200 mg BIW | Part A2: M4344 100 mg BID | Part A2: M4344 150 mg QD | Part A2: M4344 250 mg QD | Part A2: M4344 350 mg QD | Part B1: M4344 350 mg + Carboplatin | Part B1: M4344 400 mg + Carboplatin | Part B1: M4344 500 mg + Carboplatin | Part C: M4344 250 mg QD
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 1/2 | 0/1 | 1/1 | 1/2 | 1/4 | 8/12 | 3/10 | 1/7 | 5/7 | 3/5 | 2/7 | 3/7 | 1/3 | 4/7 | 2/6 | 6/13
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/1 | 1/2 | 0/1 | 1/1 | 0/2 | 2/4 | 6/12 | 6/10 | 4/7 | 5/7 | 1/5 | 2/7 | 5/7 | 1/3 | 4/7 | 3/6 | 7/13
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 1/2 | 1/1 | 1/1 | 2/2 | 4/4 | 12/12 | 10/10 | 7/7 | 7/7 | 5/5 | 7/7 | 7/7 | 3/3 | 7/7 | 6/6 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: M4344 10 mg BIW (N=2) | Part A: M4344 20 mg BIW (N=1) | Part A: M4344 40 mg BIW (N=2) | Part A: M4344 80 mg BIW (N=1) | Part A: M4344 160 mg BIW (N=1) | Part A: M4344 300 mg BIW (N=2) | Part A: M4344 450 mg BIW (N=4) | Part A: M4344 700 mg BIW (N=12) | Part A: M4344 1050 mg BIW (N=10) | Part A: M4344 1200 mg BIW (N=7) | Part A2: M4344 100 mg BID (N=7) | Part A2: M4344 150 mg QD (N=5) | Part A2: M4344 250 mg QD (N=7) | Part A2: M4344 350 mg QD (N=7) | Part B1: M4344 350 mg + Carboplatin (N=3) | Part B1: M4344 400 mg + Carboplatin (N=7) | Part B1: M4344 500 mg + Carboplatin (N=6) | Part C: M4344 250 mg QD (N=13)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Euthanasia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: M4344 10 mg BIW (N=2) | Part A: M4344 20 mg BIW (N=1) | Part A: M4344 40 mg BIW (N=2) | Part A: M4344 80 mg BIW (N=1) | Part A: M4344 160 mg BIW (N=1) | Part A: M4344 300 mg BIW (N=2) | Part A: M4344 450 mg BIW (N=4) | Part A: M4344 700 mg BIW (N=12) | Part A: M4344 1050 mg BIW (N=10) | Part A: M4344 1200 mg BIW (N=7) | Part A2: M4344 100 mg BID (N=7) | Part A2: M4344 150 mg QD (N=5) | Part A2: M4344 250 mg QD (N=7) | Part A2: M4344 350 mg QD (N=7) | Part B1: M4344 350 mg + Carboplatin (N=3) | Part B1: M4344 400 mg + Carboplatin (N=7) | Part B1: M4344 500 mg + Carboplatin (N=6) | Part C: M4344 250 mg QD (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 4 | 2 | 1 | 4 | 3 | 7
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 4 | 2 | 1 | 2 | 2 | 0 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 2 | 2 | 2 | 1 | 0 | 1 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 8 | 6 | 5 | 3 | 2 | 4 | 2 | 2 | 2 | 3 | 6
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 7 | 4 | 4 | 1 | 0 | 5 | 3 | 1 | 0 | 1 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 4 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 7 | 5 | 3 | 3 | 3 | 5 | 3 | 3 | 4 | 5 | 3
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 3 | 2 | 0 | 1 | 0 | 3
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 0 | 2 | 1 | 0 | 2 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 3
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 4 | 2 | 2 | 2 | 5 | 1 | 2 | 2 | 10
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 4 | 3 | 2 | 2 | 4 | 0 | 2 | 1 | 11
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2 | 4 | 1 | 4 | 1 | 1 | 0 | 0 | 8
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mean cell volume increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 2 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmic migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 4 | 1 | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT02278250/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT02278250/SAP_001.pdf